CLINICAL TRIAL: NCT04218539
Title: Repeat Dosing of Psilocybin in Headache Disorders
Brief Title: Repeat Dosing of Psilocybin in Migraine Headache
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: The Wallace Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2000026974; 000 (Other: CTGTY)
Record Dates: First submitted 2019-12-20; First posted 2020-01-06 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2024-02

CONDITIONS: Migraine Headache
Keywords: psilocybin; inflammation; calcitonin gene-related peptide (CGRP); pituitary adenylate cyclase-activating peptide (PACAP)
MeSH Terms: conditions — Migraine Disorders; Inflammation | interventions — Psilocybin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Placebo/Placebo (Experimental): Subjects will receive a dose of placebo, followed by a dose of placebo approximately 7 days later.
  Interventions: Drug: Placebo
- Placebo/Psilocybin (Experimental): Subjects will receive a dose of placebo, followed by a dose of psilocybin approximately 7 days later.
  Interventions: Drug: Psilocybin; Drug: Placebo
- Psilocybin/Placebo (Experimental): Subjects will receive a dose of psilocybin, followed by a dose of placebo approximately 7 days later.
  Interventions: Drug: Psilocybin; Drug: Placebo
- Psilocybin/Psilocybin (Experimental): Subjects will receive a dose of psilocybin, followed by a dose of psilocybin approximately 7 days later.
  Interventions: Drug: Psilocybin

INTERVENTIONS:
Drug: Psilocybin — 10mg Psilocybin
  Arms: Placebo/Psilocybin; Psilocybin/Placebo; Psilocybin/Psilocybin
Drug: Placebo — 25mg Diphenhydramine
  Arms: Placebo/Placebo; Placebo/Psilocybin; Psilocybin/Placebo

SUMMARY:
In seeking to understand the capacity for psilocybin to reduce migraine headache burden, this study will investigate single and repeated dosing of psilocybin up to two doses. In seeking to identify an underlying mechanism in psilocybin's effects, neuroinflammatory markers for migraine headache will be measured.

DETAILED DESCRIPTION:
Migraine headache is a common medical condition and a top cause of disability worldwide. Treatment options for migraine headache are many and varied, though an approximated 10% of migraineurs is refractory to medication and thus, there is a need to develop alternative treatments. There is anecdotal evidence supporting lasting therapeutic effects after limited dosing of psilocybin and related compounds in headache disorders. The cause of this unique effect remains unknown, though the drug class has demonstrable anti-inflammatory activity, a biological process relevant to migraine and other headache disorders. In seeking to understand the capacity for psilocybin to reduce migraine headache burden, this study will investigate single and repeated dosing of psilocybin up to two doses. In seeking to identify an underlying mechanism in psilocybin's effects, neuroinflammatory markers for migraine headache will be measured. The results from this study will serve in the development of larger investigations seeking to understand the effects of psilocybin and related compounds in headache disorders.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of migraine headache per ICHD-3 criteria
* Typical pattern of migraine attacks with approximately two migraines or more weekly
* Attacks are managed by means involving no more than twice weekly triptan use

Exclusion Criteria:

* Axis I psychotic or manic disorder (e.g., schizophrenia, bipolar I, depression with psychosis)
* Axis I psychotic or manic disorder in first degree relative
* Unstable medical condition; severe renal, cardiac, or hepatic disease; pacemaker; or serious central nervous system pathology
* Pregnant, breastfeeding, lack of adequate birth control
* History of intolerance to psilocybin, lysergic acid diethylamide (LSD), or related compounds
* Drug abuse within the past 3 months (excluding tobacco)
* Urine toxicology positive to drugs of abuse
* Alcohol use of >21 drinks per week (males); >14 drinks per week (females; NIAAA guidelines)
* Use of alcohol in the week prior to the first test day
* Use of vasoconstrictive medications (i.e., sumatriptan, pseudoephedrine, midodrine) within 5 half-lives of test days
* Use of serotonergic antiemetics (i.e., ondansetron) in the past 2 weeks
* Use of antidepressant medication (i.e., TCA, MAOI, SSRI) in the past 6 weeks
* Use of steroids or certain other immunomodulatory agents (i.e., azathioprine) in the past 2 weeks
* Use of migraine onabotulinum toxin (i.e., Botox) or monoclonal antibodies against CGRP or its receptor (i.e., erenumab) in the past month or while therapeutic effects are still present

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2021-08-10 (Actual); Primary Completion 2023-11-05 (Actual); Study Completion 2023-11-05 (Actual)

PRIMARY OUTCOMES:
Change in migraine attack frequency | From two weeks before the first session to two months after second session using a headache diary
  Average number (number per week)
Change in pain intensity of migraine attacks | From two weeks before the first session to two months after second session using a headache diary
  Average pain intensity (4-tiered pain score; 0=none, 1=mild, 2=moderate, 3=severe)
Change in duration of migraine attacks | From two weeks before the first session to two months after second session using a headache diary
  Average duration (measured in hours)
Change in intensity of photophobia (light sensitivity) | From two weeks before the first session to two months after second session using a headache diary
  Average intensity (4-tiered pain score; 0=none, 1=mild, 2=moderate, 3=severe)
Change in intensity of phonophobia (noise sensitivity) | From two weeks before the first session to two months after second session using a headache diary
  Average intensity (4-tiered pain score; 0=none, 1=mild, 2=moderate, 3=severe)
Average intensity of nausea/vomiting | From two weeks before the first session to two months after second session using a headache diary
  Average intensity (4-tiered pain score; 0=none, 1=mild, 2=moderate, 3=severe)
Change in functional disability | From two weeks before the first session to two months after second session using a headache diary
  Average disability (4-tiered pain score; 0=none, 1=mild, 2=moderate, 3=severe)

SECONDARY OUTCOMES:
Use of abortive/rescue medication | From two weeks before the first session to two months after second session using a headache diary
  number of times per week
Time to first migraine attack | From the second session until two months after second session using a headache diary
  Measured in days
Migraine attack-free time | From two weeks before the first session to two months after second session using a headache diary
  Number of 24-hour days (may be non-consecutive)
Quality of life using the Centers for Disease Control (CDC) Health-Related Quality of Life Scale: Healthy Days Symptoms Module | From two weeks before the first session to two months after second session using a headache diary
  4 questions scored 0 to 30 each; higher numbers indicate worse quality of life.
  (1) pain-related impairment, (2) mood symptoms, (3) anxiety symptoms, (4) lack of sleep. Percent change for each measure as well as total score (range 0 to 120) will be calculated
Psychedelic effects using the 5-Dimensional Altered States of Consciousness (5D-ASC) scale | Starting on the first test day until the second test day approximately one week later; taken both test days approximately 6 hours after drug administration
  94 questions scored 0 to 100 each; higher numbers indicate greater psychedelic effects. Questions address 5 dimensions: (1) Oceanic Boundlessness (score range 0-2700), (2) Dread of Ego Dissolution (score range 0-2100), (3) Visionary Restructuralization (score range 0-1800), (4) Auditory Alterations (score range 0-1600), and (5) Vigilance Reduction (score range 0-1200). Score for each dimension as well as total score (range 0 to 9400) will be measured.
Change in blood pressure- Systolic | Starting on the first test day until the second test day approximately one week later; measured both test sessions before drug administration, every 30 min in the first hour, then hourly for 4 hours or until resolution of drug effects (~6hrs after drug)
  Maximum change from baseline during each test day (mm Hg)
Change in blood pressure- Diastolic | Starting on the first test day until the second test day approximately one week later; measured both test sessions before drug administration, every 30 min in the first hour, then hourly for 4 hours or until resolution of drug effects (~6hrs after drug)
  Maximum change from baseline during each test day (mm Hg)
Change in heart rate | Starting on the first test day until the second test day approximately one week later; measured both test sessions before drug administration, every 30 min in the first hour, then hourly for 4 hours or until resolution of drug effects (~6hrs after drug)
  Maximum change from baseline during each test day (beats per minute)
Change in peripheral oxygenation | Starting on the first test day until the second test day approximately one week later; measured both test sessions before drug administration, every 30 min in the first hour, then hourly for 4 hours or until resolution of drug effects (~6hrs after drug)
  Maximum change from baseline during each test day (SpO2)
Change in peripheral calcitonin gene-related peptide (CGRP) levels | Approximately 3 months; measured at screening, on both test days (0, 2, and 4 hours after drug administration), and follow-up (~2 months after second test day)
  Change in peripheral neuropeptide levels
Change in pituitary adenylate cyclase-activating peptide (PACAP) levels | Approximately 3 months; measured at screening, on both test days (0, 2, and 4 hours after drug administration), and follow-up (~2 months after second test day)
  Change in peripheral neuropeptide levels

CONTACTS AND LOCATIONS:
Locations (1):
- VA Connecticut Healthcare System, West Haven, Connecticut, United States